CLINICAL TRIAL: NCT07038083
Title: REal-world Data of CARdiometabolic ProtEcTion
Acronym: RED-CARPET
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, Sun Yat-sen University
Other Study IDs: RED-CARPET Study
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cardiometabolic Diseases
Keywords: Cardiometabolic Diseases; all-cause mortality; Cardiovascular death; Major adverse cardiovascular events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single-center, historical prospective cohort study including patients diagnosed with metabolic cardiovascular disease, including hypertension, diabetes, obesity, dyslipidemia, hyperuricemia. The primary outcome of the study is all-cause death and cardiovascular death, and the secondary outcome is major adverse cardiovascular events. We aim to measure associations of established or suspected cardiometabolic disease (CMD) risk factors and cardiovascular disease outcomes in a real-world representative cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Patients with clinical diagnosis of metabolic cardiovascular disease, including hypertension, diabetes, obesity, dyslipidemia, hyperuricemia.

  1. Hypertension and normal high blood pressure: Three standardized blood pressure measurements in the clinic on different days, and all the blood pressure values of the three measurements were systolic blood pressure ≥ 120 mmHg and/or diastolic blood pressure ≥ 80 mmHg;
  2. Diabetes: ① Typical symptoms of diabetes, and any of the following: ② Random blood glucose ≥ 11.1 mmol/L; ③ Fasting blood glucose (FPG) ≥ 7.0 mmol/L; ④ OGTT 2-hour postprandial blood glucose ≥ 11.1 mmol/L; ⑤ HbA1c ≥ 6.5%;
  3. Obesity and overweight: Body mass index (BMI) ≥ 24 kg/m²;
  4. Dyslipidemia: At least one of the following lipid indicators is abnormal: ① Total cholesterol (TC) ≥ 6.2 mmol/L; ② Low-density lipoprotein cholesterol (LDL-C) ≥ 4.1 mmol/L; ③ High-density lipoprotein cholesterol (HDL-C) < 1.0 mmol/L; ④ Triglyceride (TG) ≥ 2.3 mmol/L; ⑤ Lipoprotein(a) ≥ 30 mg/dL;
  5. Hyperuricemia: The fasting blood uric acid levels on two different days were > 420 μmol/L (7 mg/dL) in men and > 360 μmol/L (6 mg/dL) in women.

Exclusion Criteria:

* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with cardiometabolic diseases during hospitalization were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2044-01-01 (Estimated); Study Completion 2044-01-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | Through study completion, an average of 5 years
  Death due to any cause after enrollment
Cardiovascular death | Through study completion, an average of 5 years
  Death caused by cardiac causes

SECONDARY OUTCOMES:
Major adverse cardiovascular events | Through study completion, an average of 5 years
  Including heart failure hospitalization, coronary heart disease, stroke, arrhythmia, valvular heart disease, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen Univerity, Guangzhou, Guangdong, China